CLINICAL TRIAL: NCT06987591
Title: Impact of Low-Dose Epidural Analgesia on Labour Progression in Robson Class 1 Women: a Retrospective Study
Brief Title: Impact of Low-Dose Epidural Analgesia on Labour Progression in Low-Risk Women
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, ZANFINI BRUNO ANTONIO, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6077
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Epidural Analgesia, Obstetric
Keywords: Labor epidural analgesia; Cesarean section; Instrumental delivery; Neonatal well-being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- VD-e: Women who vaginally delivered and received EA for labour.
- VD-n: Women who vaginally delivered and did not receive EA for labour.
- CD-e: Women who delivered via intrapartum caesarean section and received EA for labour.
- CD-n: Women who delivered via intrapartum caesarean section and did not receive EA for labour.

SUMMARY:
Aim of the study was to analyse data on cervical dilation and fetal descent patterns in low-risk women, who did or did not receive intermittent low-dose epidural analgesia (EA), and who had either a vaginal or a caesarean delivery.

Therefore, we conducted a retrospective analysis, retrieving data from October 1st 2008 to October 31st 2018. We selected 6030 women categorized as Robson Group 1, divided into four groups according to the mode of delivery (vaginal or caesarean) and the presence of EA:

* Vaginal delivery with EA (VD-e)
* Vaginal delivery without EA (VD-n)
* Caesarean delivery with EA (CD-e)
* Caesarean delivery without EA (CD-n)

ELIGIBILITY:
Inclusion Criteria:

* Robson class 1 (nulliparous, single, cephalic full-term pregnancy with spontaneous labour)
* maternal age between 18 and 40 years
* neonatal weight between 2500 and 4000 grams
* cervical dilation <7 cm at admission in the delivery suite

Exclusion Criteria:

* minimal duration of labour < 3 hours (from admission to the delivery suite to delivery)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant patients classified as Robson class 1, who received or not EA for labour and delivered either vaginally or via caesarean route.
Sampling Method: Non-Probability Sample
Enrollment: 5995 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Cervical dilation curve | First stage of labour (from admission to the delivery suite to full cervical dilation)
  We modeled the cervical dilation curve using a high-degree mixed polynomial regression. The analysis was conducted separately in women with vaginal or caesarean delivery. The time of complete cervical dilation or caesarean delivery was considered the point 0 for cervical dilation, while the preceding events resulted in negative time compared to the 0.
Fetal head descent curve | From admission to the delivery room up to the time of delivery (either via vaginal route or caesarean section)
  We modeled the fetal head descent curve using a mixed polynomial regression. The analysis was conducted separately in women with vaginal or caesarean delivery. The time of station +3 (i.e. vaginal birth) or caesarean delivery was considered the point 0 , while the preceding events resulted in negative time compared to the 0.

SECONDARY OUTCOMES:
Length of active phase | Up to 24 hours from admission.
  The beginning of the active phase was defined in the presence of regular painful uterine contractions, a substantial degree of cervical effacement and more rapid cervical dilation. Active phase ends at full cervical dilation.
Length of second stage | Up to 24 hours from admission.
  Second stage begins at full cervical dilation and ends at delivery.
Type of vaginal delivery | At delivery
  In the VD-e and VD-n groups, description of the type of delivery (eutocic or instrumental)
Maternal complications during vaginal delivery | At delivery.
  Rate of maternal complications (postpartum haemorrhages, perineal lacerations, uterine atony) in the VD groups.
Episiotomy | At delivery.
  Rate of episiotomy in the VD groups.
Fetal indicators | After delivery
  Apgar at 1 and 5 minutes, admission in Neonatal Intensive Care Unit (NICU), death

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No
For patient's privacy protection.

REFERENCES:
- [Background] Anim-Somuah M, Smyth RM, Cyna AM, Cuthbert A. Epidural versus non-epidural or no analgesia for pain management in labour. Cochrane Database Syst Rev. 2018 May 21;5(5):CD000331. doi: 10.1002/14651858.CD000331.pub4. PMID 29781504
- [Background] de Vries BS, Mcdonald S, Joseph FA, Morton R, Hyett JA, Phipps H, McGeechan K. Impact of analysis technique on our understanding of the natural history of labour: a simulation study. BJOG. 2021 Oct;128(11):1833-1842. doi: 10.1111/1471-0528.16719. Epub 2021 May 19. PMID 33837643
- [Background] Vahratian A, Troendle JF, Siega-Riz AM, Zhang J. Methodological challenges in studying labour progression in contemporary practice. Paediatr Perinat Epidemiol. 2006 Jan;20(1):72-8. doi: 10.1111/j.1365-3016.2006.00696.x. PMID 16420344
- [Background] Friedman EA. Evolution of graphic analysis of labor. Am J Obstet Gynecol. 1978 Dec 1;132(7):824-7. doi: 10.1016/s0002-9378(78)80018-0. No abstract available. PMID 717493
- [Background] Zhang J, Troendle JF, Yancey MK. Reassessing the labor curve in nulliparous women. Am J Obstet Gynecol. 2002 Oct;187(4):824-8. doi: 10.1067/mob.2002.127142. PMID 12388957
- [Background] Zhang J, Landy HJ, Ware Branch D, Burkman R, Haberman S, Gregory KD, Hatjis CG, Ramirez MM, Bailit JL, Gonzalez-Quintero VH, Hibbard JU, Hoffman MK, Kominiarek M, Learman LA, Van Veldhuisen P, Troendle J, Reddy UM; Consortium on Safe Labor. Contemporary patterns of spontaneous labor with normal neonatal outcomes. Obstet Gynecol. 2010 Dec;116(6):1281-1287. doi: 10.1097/AOG.0b013e3181fdef6e. PMID 21099592